CLINICAL TRIAL: NCT07315971
Title: The Effect Of Health Development Behavıour Traınıng In Pregnancy On Sleep Qualıty And Physıcal Actıvıty Levels: A Randomızed Controlled Experımental Study
Brief Title: The Effect Of Health Development Behavıour Traınıng In Pregnancyon Sleep Qualıty And Physıcal Actıvıty Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Fatma Kurt, Dr. Ph.D., Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-21347915-050.04.04-264603l; Randomızed Controlled Experıme (Registry Identifier: Randomızed Controlled Experıme)
Record Dates: First submitted 2025-11-20; First posted 2026-01-05 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Health Behavior; Physical Activity; Sleep Quality
Keywords: Exercise; Education; Pregnancy; Nursing; Sleep
MeSH Terms: conditions — Health Behavior; Motor Activity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Following recruitment, the pregnant women were divided into a study and a control group by randomization (1:2 randomization)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The study group received training on health promotion during pregnancy in addition to usual care provided by health professionals.
  Interventions: Behavioral: HEALTH PROMOTION BEHAVIOR TRAINING
- Control group (No Intervention): The control group continued to receive the routine care

INTERVENTIONS:
Behavioral: HEALTH PROMOTION BEHAVIOR TRAINING — Exercise During Pregnancy When Should Exercise Be Started During Pregnancy? Which Exercises Are Recommended/Not Recommended During Pregnancy? How Intense Should Exercise Be During Pregnancy? How Long Should Exercise Last? Points to Consider When Exercising Exercise Examples Health Responsibility Pregnancy Monitoring Smoking During Pregnancy, Alcohol, and Substance Use During Pregnancy Sexuality During Pregnancy Hygiene and General Care During Pregnancy Sleep During Pregnancy Sleep Problems During Pregnancy Recommendations for Quality Sleep During Pregnancy Interpersonal Relationships Effective Communication Skills Stress Management Factors That Can Cause Stress During Pregnancy Positive Methods for Coping with Stress During Pregnancy The intervention group received 6 weeks of face-to-face training.
  Arms: experimental group

SUMMARY:
The aim of this study is to determine the effect of health-promoting behavior education on the sleep quality and physical activity levels of pregnant women. 1.2. The research hypotheses are as follows:

H0 hypotheses:

* Ho (1): Education on healthy lifestyle behaviors during pregnancy does not affect sleep quality in pregnant women.
* Ho (2): Education on healthy lifestyle behaviors during pregnancy does not affect physical activity levels in pregnant women.

H1 hypotheses:

* H1 (1): Education on healthy lifestyle behaviors during pregnancy improves sleep quality in pregnant women.
* H1 (2): Education on healthy lifestyle behaviors during pregnancy increases physical activity levels in pregnant women.

The study group received health promotion training for six weeks. Data were collected by administering the scales three times: before, immediately after, and one month later. The control group received no training and only underwent routine pregnancy examinations and follow-up at the family health center. The scales were administered at the same times as the pregnant women in the study group.

DETAILED DESCRIPTION:
This study is a pre-test post-test randomized controlled experimental research. The population of the study consisted of 620 pregnant women, and the sample included a total of 57 pregnant women, with 27 in the experimental group and 30 in the control group. Prior to the intervention, individual interviews were conducted, and written consent was obtained from the participants. Subsequently, the questionnaire prepared by the researcher, the Pittsburgh Sleep Quality Index (PSQI), and the Pregnancy Physical Activity Questionnaire (PPAQ) were administered. The experimental group received health-promoting behavior education for six weeks, with sessions held once a week for 30 minutes at a Family Health Center, in a room designated by the center's staff during working hours. At the end of the training, the scales were administered again, and one month after the completion of the education, the PSQI and PPAQ were re-administered. The data obtained from the study were analyzed using the SPSS 25.0 package program at a 95% confidence interval and a significance level of 0.05. The normal distribution of the data was evaluated using the Kolmogorov-Smirnov test. Parametric tests were used when normal distribution assumptions were met, and non-parametric tests were applied when these assumptions were not satisfied.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who were: • in the early third trimester,

  * had at least a primary school education,
  * had no communication barriers were included.

Exclusion Criteria:

Incomplete completion of the data collection tools used in the study,

* Having a psychiatric diagnosis (major depression, psychotic disorders, intellectual disability),
* Being pregnant under the age of 18,
* Having a chronic disease (such as diabetes, heart disease, hypertension, cancer),
* Multiple pregnancy were considered exclusion criteria.
* Not following the training programs included in the study (at least two trainings),

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 57 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Physical Activity Questionnaire for Pregnant Women | 28th week of pregnancy
  Physical Activity Questionnaire for Pregnant WomenThe Turkish validity and reliability of the scale, developed by Chasan Taber et al. in 2004, was determined by Çırak et al. It consists of 36 questions that determine the level of physical activity and exercise in pregnant women. This scale evaluates 32 activities performed by pregnant women: housework and care activities (n=13), occupational activities (n=5), sports and exercise activities (n=8), transportation (n=3), and sedentary lifestyle (n=3). The intensity of physical activity is expressed in METs (metabolic equivalents). In open-ended questions, the MET value of the activity is determined by referring to the Review. Activity intensities are grouped as sedentary (0.6 MET). Activity types are classified as housework/care activities, occupational activities, and sports/exercise. In this study, the Cronbach's alpha coefficient of the scale was found to be 0.65.
The Pittsburgh Sleep Quality Index | 28th week of pregnancy
  PSQI developed by Buysse et al. has been shown to have sufficient internal consistency (Cronbach's alpha = 0.80), test-retest reliability, and validity (Buysse et al. It was adapted into Turkish by Ağargün et al. The PSQI is a 19-item self-report scale that assesses sleep quality and disturbance over the past month. It consists of 24 questions: 19 self-report questions and 5 questions to be answered by a spouse or roommate. The 18 scored questions comprise 7 components: Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disturbance, Sleep Medication Use, and Daytime Dysfunction. Each component is scored on a scale of 0-3. The total score of the 7 components gives the total scale score. The total score ranges from 0-21. A total score greater than 5 indicates "poor sleep quality". Permission was obtained for the scale's use. Cronbach's alpha coefficient of the scale was found to be 0.71.

SECONDARY OUTCOMES:
Physical Activity Questionnaire for Pregnant Women | 33th week of pregnancy
  The Turkish validity and reliability of the scale, developed by Chasan Taber et al. in 2004, was determined by Çırak et al. It consists of 36 questions that determine the level of physical activity and exercise in pregnant women. This scale evaluates 32 activities performed by pregnant women: housework and care activities (n=13), occupational activities (n=5), sports and exercise activities (n=8), transportation (n=3), and sedentary lifestyle (n=3). The intensity of physical activity is expressed in METs (metabolic equivalents). In open-ended questions, the MET value of the activity is determined by referring to the Review. Activity intensities are grouped as sedentary (0.6 MET). Activity types are classified as housework/care activities, occupational activities, and sports/exercise. In this study, the Cronbach's alpha coefficient of the scale was found to be 0.65.
The Pittsburgh Sleep Quality Index | 33th week of pregnancy
  PSQI developed by Buysse et al. has been shown to have sufficient internal consistency (Cronbach's alpha = 0.80), test-retest reliability, and validity. It was adapted into Turkish by Ağargün et al. The PSQI is a 19-item self-report scale that assesses sleep quality and disturbance over the past month. It consists of 24 questions: 19 self-report questions and 5 questions to be answered by a spouse or roommate. The 18 scored questions comprise 7 components: Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disturbance, Sleep Medication Use, and Daytime Dysfunction. Each component is scored on a scale of 0-3. The total score of the 7 components gives the total scale score. The total score ranges from 0-21. A total score greater than 5 indicates "poor sleep quality". Permission was obtained for the scale's use. Cronbach's alpha coefficient of the scale was found to be 0.71.

OTHER OUTCOMES:
Physical Activity Questionnaire for Pregnant Women | 38th gestational weeks
  The Turkish validity and reliability of the scale, developed by Chasan Taber et al. in 2004, was determined by Çırak et al. It consists of 36 questions that determine the level of physical activity and exercise in pregnant women. This scale evaluates 32 activities performed by pregnant women: housework and care activities (n=13), occupational activities (n=5), sports and exercise activities (n=8), transportation (n=3), and sedentary lifestyle (n=3). The intensity of physical activity is expressed in METs (metabolic equivalents). In open-ended questions, the MET value of the activity is determined by referring to the Review. Activity intensities are grouped as sedentary (0.6 MET). Activity types are classified as housework/care activities, occupational activities, and sports/exercise. In this study, the Cronbach's alpha coefficient of the scale was found to be 0.65.
The Pittsburgh Sleep Quality Index | 38th gestational weeks
  PSQI developed by Buysse et al. has been shown to have sufficient internal consistency (Cronbach's alpha = 0.80), test-retest reliability, and validity. It was adapted into Turkish by Ağargün et al. The PSQI is a 19-item self-report scale that assesses sleep quality and disturbance over the past month. It consists of 24 questions: 19 self-report questions and 5 questions to be answered by a spouse or roommate. The 18 scored questions comprise 7 components: Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disturbance, Sleep Medication Use, and Daytime Dysfunction. Each component is scored on a scale of 0-3. The total score of the 7 components gives the total scale score. The total score ranges from 0-21. A total score greater than 5 indicates "poor sleep quality". Permission was obtained for the scale's use. Cronbach's alpha coefficient of the scale was found to be 0.71.

CONTACTS AND LOCATIONS:
Overall Officials: Safiye Özvurmaz, Phd, Study Director — Aydın Adnan Menderes University, Faculy of Nursing, Division Public Health Nursing
Locations (1):
- Aydın Adnan Menderes Üniversitesi, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.